CLINICAL TRIAL: NCT06971562
Title: Effect of Silver on Re-epithelialization, Infection and Hypertrophic Scarring of Partial Thickness Burns in Pediatric Patients: A Randomized Controlled Trial
Brief Title: Silver in Partial Thickness Pediatric Burns
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Michael Bezuhly, Principal Investigator, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1022040
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Pediatric Burns
Keywords: silver; burn dressing; re-epithelialization; scarring; infection
MeSH Terms: conditions — Cicatrix; Infections

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquacel (Active Comparator): Aquacel hydrocellulose-based dressing applied to partial thickness burns
  Interventions: Device: Aquacel
- Aquacel AG (Active Comparator): Aquacel AG is identical in base composition to Aquacel (ie a hydrocellulose-based wound dressing which adheres to the raw wound surface) but contains 1.2% cationic silver.
  Interventions: Device: Aquacel AG

INTERVENTIONS:
Device: Aquacel AG — Hydrocellulose wound dressing containing 1.2% cationic silver
  Arms: Aquacel AG
Device: Aquacel — Hydrocellulose wound dressing
  Arms: Aquacel

SUMMARY:
Most burns in children are due to scalds and with proper dressings will heal on their own without the need for surgery such as skin grafting. Many current burn dressings contain silver which is felt to reduce the risk of infection. Unfortunately, when applied to burns, silver causes pain and may actually slow healing. The aim of this study is to compare the time it takes for less severe burns in children to heal when they are treated with two forms of the same dressing, one that contains silver and another that does not. In addition, we will check to see if there is a difference between dressings in terms of the risk of infection and the quality of the healed skin.

DETAILED DESCRIPTION:
This randomized controlled single-blind trial will examine the effect of silver in dressings to healing of superficial partial thickness burns in a pediatric population. Briefly, patients under the age of 16 with <25% total body surface area (TBSA) superficial partial thickness burns not exclusively to the perineum, face, hands, or feet, no inhalational, chemical or electrical burns and no other concomitant injuries presenting to the plastic surgery service < 72 hours after injury will be eligible to receive a hydrocellulose dressing either without (Aquacel) or with silver (Aquacel AG) to their burns. Patients will be excluded if they have a documented allergy to silver. Demographic and clinical information (including mechanism of injury and area involved) will be collected after informed consent is obtained. Photographs and surface area of the burned area will be recorded using an app (LesionMeter, version 1.1). Using a computer generated block randomization sequence, patients will either have Aquacel or Aquacel AG applied to their burn by a burn nurse. Patients then follow-up in clinic 7-10 days later to assess the extent of re-epithelialization. As the Aquacel dressing separates from skin once it has re-epithelialized, the extent of non-healed burn will be assessed by the plastic surgeon blinded to the patient's treatment group by assessing the amount of dressing still adherent once it has been trimmed. Follow-up is then performed every two days after the initial dressing until the dressing has completely separated. Subsequent follow-up visits are then performed at 3 and 6 months after injury during which a Vancouver Scar Scale assessment is performed by an occupational therapist blinded to the treatment group of the patient. The primary outcome will be time-to-re-epithelialization in days, with secondary outcomes including rate of infection per treatment group and difference in mean Vancouver Scar Scale scores at 3- and 6-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* <16 years old
* partial thickness thermal (scald, contact, fire) burns up to 25% TBSA on the trunk and extremities
* presenting < 72 hours after injury

Exclusion Criteria:

* mixed burn pattern (combination of partial and full thickness burn) or full thickness burns requiring surgery at either anatomic sites.
* isolated burns to perineum, hands, or feet allergy to silver
* concomitant injury (eg.fractures)
* inhalational injury
* chemical burn
* electrical burn
* unable to understand English or French
* have not had a silver-based wound dressing applied prior to presentation

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Time-to-re-epithelialization | 10-21 days
  Time (in days) for complete re-epithelialization of the burn to which the dressing was applied

SECONDARY OUTCOMES:
Rate of infection | 3 months
  Incidence of infection in each study arm
Vancouver Scar Scale (VSS) score | 3 and 6 months post-injury
  Mean cumulative VSS score for each Arm.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bezuhly, MD, MSc, SM, FRCSC, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided